CLINICAL TRIAL: NCT05064696
Title: Prospective Comparison of Wound Complications After Anterior Total Ankle Arthroplasty With and Without PICO Negative Pressure Incisional Dressing
Brief Title: PICO- Single-use Negative Pressure Wound Therapy System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter C Hembree (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Walter C Hembree, MD, Medstar Health Research Institute
Organization: Medstar Health Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003790
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Total Ankle Arthroplasty
Keywords: Total ankle arthroplasty; PICO; Ankle; Ankle joint; Arthroplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Control group) (Active Comparator): Surgical wound will be covered with the standard non-stick gauze dressing.
  Interventions: Other: Non-stick gauze dressing
- Group 2 (Treatment group) (Experimental): Surgical wound will be covered with the PICO dressing.
  Interventions: Device: PICO dressing

INTERVENTIONS:
Other: Non-stick gauze dressing — Group 1 (Control group): surgical site will be dressed with a standard non-stick gauze dressing
  Arms: Group 1 (Control group)
Device: PICO dressing — Group 2 (Treatment group): surgical site will be dressed with PICO dressing
  Arms: Group 2 (Treatment group)

SUMMARY:
To compare the rate of wound complications with the PICO dressing versus a standard nonstick gauze dressing in patients undergoing anterior total ankle arthroplasty.

DETAILED DESCRIPTION:
Participating subjects will be randomized to one of the study groups: Group 1 (Control group) or Group 2 (Treatment group). If randomized to Group 1- after surgery, the doctor will apply the standard non-stick gauze dressing to the wound. If randomized to Group 2- after surgery, the doctor will apply the PICO dressing to the wound.

The goal of the study is to measure the rate of wound complications based on wound assessment, patient-reported outcomes surveys, as well as peri- and post-operative data.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old
* Subjects undergoing total ankle arthroplasty or uncomplicated revision total ankle arthroplasty
* Subjects able to provide informed consent
* Subjects who are able to understand and comply with study visit schedule and procedures

Exclusion Criteria:

* History of previous deep infection or history of wound complication necessitating plastic surgery intervention
* Allergy to products used in the study
* Pregnant and breastfeeding women due to anesthesia risks
* Subjects with a known history of poor compliance with medical treatment
* Subjects who decline participation in this research study
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Wound complications | Approximately 12-weeks after surgery (or until 3-month postop visit is completed)
  To determine presence or absence of wound complications at the follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Walter C Hembree, MD, Principal Investigator — MedStar Health
Locations (1):
- Amy Loveland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No